CLINICAL TRIAL: NCT00539708
Title: Non-Invasive Ventilation After Extubation in Hypercapnic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Fondo de Investigacion Sanitaria (Other)
Responsible Party: Miquel Ferrer, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FIS 041130
Record Dates: First submitted 2007-10-03; First posted 2007-10-04 (Estimated); Last update posted 2008-05-12 (Estimated); Status verified 2008-05

CONDITIONS: Respiratory Failure
Keywords: Non-invasive ventilation; Hypercapnic respiratory failure; Mechanical ventilation; Respiratory failure after extubation
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NIV (Experimental): Non-invasive ventilation
  Interventions: Procedure: Non-invasive ventilation
- Control (Active Comparator): Oxygen therapy
  Interventions: Procedure: Non-invasive ventilation

INTERVENTIONS:
Procedure: Non-invasive ventilation — Non-invasive ventilation after extubation for 24 hours

SUMMARY:
The purpose of this study is to assess the efficacy of noninvasive ventilation in the prevention of extubation failure and mortality in patients with chronic respiratory disorders and hypercapnic respiratory failure during spontaneous breathing.

DETAILED DESCRIPTION:
Background and aims: Patients with chronic respiratory disorders, intubated and mechanically-ventilated in intensive care units (ICU), often exhibit hypercapnia during the spontaneous breathing trial prior to extubation; this is associated to increased incidence of extubation failure and mortality. We will assess the efficacy of noninvasive ventilation (NIV) in the prevention of extubation failure and mortality in these patients. Design: Prospective, randomized, controlled clinical trial with two groups: support with noninvasive ventilation, and conventional clinical management (control group). Subjects: Patients with chronic respiratory disorders, intubated and ventilated ³48 hours, with hypercapnia (PaCO2 >45 mmHg) during the spontaneous breathing trial, ready to be extubated. Interventions: Random allocation into two groups: NIV immediately after extubation during 24 hours, on conventional clinical management. Clinical follow-up (incidence of extubation failure, reintubation, ICU and hospital mortality, 90-day survival, complications associated to mechanical ventilation, ICU and hospital length of stay). Analyses of data: Comparison between two groups (NIV and control) in non-paired data design: quantitative variables (t-test, Mann-Whitney test, ROC curves), qualitative or categorical variables (chi square, Fisher's exact test), and Kaplan-Meier estimate of survival curves).

ELIGIBILITY:
Inclusion Criteria:

* Chronic respiratory disorders with invasive mechanical ventilation
* Hypercapnic respiratory failure during successful spontaneous breathing trial

Exclusion Criteria:

* Face or cranial trauma or surgery
* Recent gastric or esophageal surgery
* Tracheostomy or other upper airway disorders
* Upper gastrointestinal bleeding
* Excess respiratory secretions
* Lack of collaboration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2005-05; Primary Completion 2008-01 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Primary outcome: The incidence of respiratory failure after extubation | 3 days after extubation

SECONDARY OUTCOMES:
Survival | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Miquel Ferrer, MD, PhD, Principal Investigator — UVIIR. Servei de Pneumologia, Hospital Clinic,Barcelona
Locations (1):
- Hospital Clinic, Barcelona, Spain

REFERENCES:
- [Derived] Ferrer M, Sellares J, Valencia M, Carrillo A, Gonzalez G, Badia JR, Nicolas JM, Torres A. Non-invasive ventilation after extubation in hypercapnic patients with chronic respiratory disorders: randomised controlled trial. Lancet. 2009 Sep 26;374(9695):1082-8. doi: 10.1016/S0140-6736(09)61038-2. Epub 2009 Aug 12. PMID 19682735